CLINICAL TRIAL: NCT05626062
Title: Toileting Assessment and Toilet Training for Adults With Learning Disabilities With Incontinence
Brief Title: Toilet Training and Adults With Learning Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glasgow Caledonian University (Other)
Collaborators: University of Kent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R4451
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Urinary Incontinence
Keywords: Incontinence; Learning disabilities
MeSH Terms: conditions — Urinary Incontinence; Learning Disabilities

STUDY DESIGN:
Intervention Model Description: A feasibility sample of 30 adults with learning disabilities with incontinence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): 30 adults with learning disabilities with incontinence will be offered a 12-week personalised toilet training plan, which promotes prompted voiding in a toilet
  Interventions: Device: Toilet alarm

INTERVENTIONS:
Device: Toilet alarm — A Malem toilet alarm (wristworn, discretely in underwear, or bed mat) will be used to promote prompred voiding in a toilet

SUMMARY:
Incontinence is common in adults with learning disabilities (LDs). Behavioural toilet training in conjunction with toilet alarms is recommended for people with LDs, but there is a paucity of research, thus evidence-based practise, on behavioural toilet training for adults with LDs. The aim of this study is to assess the toileting needs and issues of 30 adults with LDs with incontinence, and determine whether a 12-week individualised positive behavioural support training intervention, with the use of toilet alarms, promotes continence.

DETAILED DESCRIPTION:
Adults with learning disabilities with incontinence are being invited to participate in a 12-week personalised, positive toilet training plan, following assessment of their toileting needs. Primary outcome measures will be: number of incidences of incontinence, and number of instances of successful voiding in a toilet. Toilet alarms will be used to encourage prompted voiding in a toilet.

ELIGIBILITY:
Inclusion Criteria:

- Adults with learning disabilities with incontince across all levels of learning disabilities (mild to profound)

Exclusion Criteria:

* Cannot sit on a toilet for up to 3 minutes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-28 (Actual); Primary Completion 2023-09-27 (Estimated); Study Completion 2023-11-27 (Estimated)

PRIMARY OUTCOMES:
Number of instances of incontinence | 12 weeks
  The intervention should promote less instances of incontinence
Number of instances of successful voiding in a toilet | 12 weeks
  The intervention should promote more instances of successful voiding in a toilet

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Glasgow Caledonian University, Glasgow, Lanarkshire
  - Glasgow Caledonian University, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finlayson J, Gore N, Ord P, Roche F, Butcher J, Kean R, Skelton DA. Urinary Tract Infections Amongst Adults With Intellectual Disabilities With Urinary Incontinence. J Appl Res Intellect Disabil. 2025 Jan;38(1):e13317. doi: 10.1111/jar.13317. PMID 39508283